CLINICAL TRIAL: NCT06275451
Title: Qualitative Study of Emotional Regulation in Schizophrenia
Acronym: QUALI-RES
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: EssaiClinique_QUALI-RES
Record Dates: First submitted 2024-01-31; First posted 2024-02-23 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia; Schizophrenia Schizoaffective
Keywords: Psychosis; Qualitative study
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Semi-structured interview: Semi-structured interview
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — Semi-structured interview on emotional regulation and administration of questionnaires lasting approximately 2 hours.

SUMMARY:
The main aim of this study is to investigate emotional regulation in individuals with schizophrenia using a qualitative methodology (semi-structured interview) and, therefore, from the person's point of view.

Given the qualitative nature of the methodology used in this study, the investigators have no specific hypothesis. The investigators have a general hypothesis suggesting that the patients' discourse will enable us to highlight the emotional regulation difficulties described in the literature.

DETAILED DESCRIPTION:
Emotional regulation (ER) is conceptualised as a transdiagnostic process involved in the development and maintenance of various mental disorders. Emotion regulation strategies have traditionally been classified as maladaptive or adaptive. Adapted emotion regulation strategies are thought to protect against psychopathology, whereas maladaptive strategies are considered to be psychopathological risk factors.However, recent theoretical models indicate that strategy choices need to be studied in relation to context and the notion of flexibility in emotional regulation. The notion of flexibility in emotional regulation refers to the individual's ability to use a repertoire of ER strategies to manage emotions according to contextual demands.The role of emotional dysregulation in psychotic disorders has emerged as a consubstantial feature of psychosis with important implications for its onset and maintenance. Individuals suffering from a psychotic disorder or reporting psychotic-like experiences (PLEs) have great difficulty regulating their emotions effectively. However, knowledge about emotional regulation in psychosis has been predominantly quantitative, neglecting patients' own perceptions.

The main aim of this study is to investigate emotional regulation in individuals with schizophrenia using a qualitative methodology (semi-structured interview) and, therefore, from the person's point of view.

Secondary objectives:

1. To study the stages of emotional regulation in individuals suffering from schizophrenia using a qualitative methodology (semi-structured interview) in line with theoretical models in psychology.
2. To study the factors that appear to influence emotional regulation in individuals with schizophrenia using a qualitative methodology (semi-structured interview) and, therefore, from the person's point of view.
3. To study, from the person's point of view, what could be useful to improve emotional regulation in individuals with schizophrenia using a qualitative methodology (semi-structured interview).

This is a type 3 study under the Jardé law, multicentre, involving the human person. This qualitative cross-sectional study includes patients diagnosed with schizophrenia from the Centre Hospitalière Alpes Isère, the Centre Hospitalière Universitaire de Grenoble Alpes and patients recruited via social networks. Its cross-sectional nature will enable us to collect data using a semi-structured interview developed specifically to explore issues relating to emotional regulation.

This study presents negligible risks or constraints for patients. The interview is designed to respect patients' time and leave them free to talk about their difficulties with emotional regulation as they wish. A large number of studies using qualitative methodology to address a range of different subjects have already demonstrated the feasibility and adaptability of these measures with patients with schizophrenia. However, these patients may find the interview tiring. To mitigate this potential risk, the investigators decided to offer an 'on-demand' interview to the subjects of the study, i.e. they will be able to complete the information form consecutively or in instalments and to take regular breaks during the interview. The interviews will be conducted by a clinical psychologist with experience of working with people with schizophrenia. Despite the possible minor risks (e.g. fatigue, discomfort) associated with this research, the investigators hope that it will lead to a better understanding of the factors involved in emotional regulation in patients with schizophrenia. Ultimately, this knowledge could lead to the development of quantitative studies to test the hypotheses that will emerge from this large-scale study and, potentially, to psychological treatments aimed at improving emotional regulation in patients with schizophrenia.

Description of the study process :

Selection visit: The selection visit will take place either during an appointment with the investigator as part of the treatment, or remotely (Zoom platform). The selection visit will be remote, particularly if the patient was recruited via social networks. For the latter, the information note will be accessible in the announcement of the study before any contact is made.

For participants followed up in the centres involved in this research, before the patient is contacted, the presence of the inclusion criteria and the absence of the study's non-inclusion criteria will be checked. For participants recruited online, during this visit the investigator will check the inclusion and non-inclusion criteria without collecting this information and/or noting it on the CRF.

The study will be presented to the patient, along with its risks and benefits, and an information letter will be provided.

Inclusion visit and Visit 1: During the inclusion visit, which is carried out either face-to-face at the next appointment with the investigator or remotely (Zoom platform), depending on the patient's preferences, the investigator will put in place arrangements to prove that the person who is to take part in the research has been informed. The investigator will also ascertain that the patient does not object to taking part in the study. The investigator will also record the patient's eligibility in the CRF.

Patients will then complete the semi-structured interview (see appendix) and fill in a General Information Form, and the CRF will be completed.

Coding methodology :

The mean and standard deviation will be calculated for all scales. For categorical variables (e.g. gender), the investigators will calculate the N and the percentage.

The data will be saved on the Université Grenoble Alpes server for the duration of the research. They will then be deleted from the university server and saved on the CHUGA servers.

The transcribed data will be read and re-read to ensure familiarity with the data. All interviews will be coded by the psychologist who conducted the interview (Emma Rolland Carlichi), but in line with recommendations, multiple coding of a number of interviews, review of the coding framework by the team (Catherine Bortolon, Céline Baeyens and Clément Dondé) and regular consultation with the team, including in the event of uncertainty during coding, will aim to increase reliability.

Two preliminary transcripts will be examined in their entirety by two members of the research team (Emma Rolland-Carlichi and Catherine Bortolon) who will each have independently recorded ideas for possible codes before discussing them. The suggested codes will then be discussed with a third member of the team (Céline Baeyens) who will also examine these initial transcriptions. A preliminary coding framework, which will therefore incorporate multiple perspectives on the data, will then be agreed. This framework will largely correspond to the main themes of the interview guide, but it may evolve as ideas emerge throughout the interviews.

The details of each code (including the specific data and coder behind the code, and whether it was an a priori or 'in vivo' code) will be recorded using memos in Nvivo, to form a codebook. The coding framework will be regularly reviewed by the research team and adjusted accordingly.

As the coding framework evolves, previous interviews will be reviewed to ensure that information relevant to emerging codes has been captured. Once all interviews have been completed, 'coding checks' will be carried out for each transcript. This will involve the lead coder reviewing their initial codes with 'fresh eyes' after a period of time, which has been recommended as a strategy to mitigate the distorting effects that immersion in the data can cause.

The interviews will be explored using inductive and deductive thematic analysis. As indicated, this approach will be used to generate initial codes, which will be constantly compared and modiﬁed as new interviews are added and analysed.

NvVivo will be used to facilitate the coding, organisation and analysis of the data.

Results:

The results of this project will initially increase our knowledge of ER in patients with schizophrenia. They will enrich the scientific literature and the theoretical models of ER applied to understanding the difficulties reported by clinical populations. In addition, the use of a qualitative method will provide ecological information on the factors involved in emotional regulation. Finally, the data obtained in this study will serve as a basis for the development of quantitative studies enabling the ER to be assessed in a more appropriate way on a large scale. Secondly, our results could guide the development of interventions targeting the use of adaptive emotional regulation strategies in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or schizoaffective disorder verified using the criteria of the M.I.N.I. (Mini International Neuropsychiatric Interview) scale (First, Spitzer, Gibbon, Williams, & others, 1995) based on the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) (Association & others, 2013).
* Patient in free care, under psychiatric care at the request of a third party or under curatorship. In the case of patients under curatorship, the investigator will inform the curator of the participant's non-opposition and therefore of his or her participation in the research.
* Able to read, understand and speak French.
* Age ≥ 18 years and < 60 years
* Must consent to the study and be able to give oral non-opposition.

Exclusion Criteria:

* Psychological instability (i.e., Agitation or major suicidal risk on clinical examination by psychiatrist prior to study entry).
* Neurological history/comorbidity (head injury, epilepsy, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Huntington's disease, stroke).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be drawn from a clinical population diagnosed with schizophrenia, aged between 18 and 60.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Emotional regulation in schizophrenia | 2 hours per participant / 2 years for research
  Emotional regulation in schizophrenia The main objective of this study is to study emotional regulation in individuals suffering from schizophrenia using a qualitative methodology (semi-structured interview) and, therefore, from the person's point of view. Semi-structured interview; The patients' discourse and the themes emerging from this discourse in relation to emotional regulation.schizophrenia

SECONDARY OUTCOMES:
Factors influencing emotional regulation in schizophrenia | 2 hours per participant / 2 years for research
  2To study the factors that appear to influence emotional regulation in individuals with schizophrenia using a qualitative methodology (semi-structured interview) and, therefore, from the person's point of view. The patients' discourse and the themes emerging from this discourse in relation to emotional regulation.
Improved emotional regulation in schizophrenia | 2 hours per participant / 2 years for research
  3. To study, from the person's point of view, what could be useful to improve emotional regulation in individuals with schizophrenia using a qualitative methodology (semi-structured interview). The patients' discourse and the themes emerging from this discourse in relation to emotional regulation.
Stages of emotional regulation in schizophrenia | 2 hours per participant / 2 years for research
  To study the stages of emotional regulation in individuals suffering from schizophrenia using a qualitative methodology (semi-structured interview) in line with theoretical models in psychology.

CONTACTS AND LOCATIONS:
Overall Officials: Clément Dondé, Principal Investigator — University Grenoble, Hospital; Catherine Bortolon, Principal Investigator — C3R and UGA
Locations (2):
- France (2):
  - CHUGA, La Tronche
  - C3R, Saint-Martin-d'Hères

IPD SHARING:
Plan to Share IPD: No